CLINICAL TRIAL: NCT01709812
Title: A 6 Months, Randomized, Multicenter, Parallel-group, Open-label Study to Evaluate the Effect of an Individualized Patient Support Program on Treatment Satisfaction in Fingolimod-treated Patients With Relapsing-remitting Multiple Sclerosis
Brief Title: Effect of an Individualized Patient Support Program on Treatment Satisfaction in Fingolimod-treated Patients With RRMS
Acronym: STAY
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720DDE19
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Relapsing-remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Standard of Care

ARMS (2):
- 1 standard care (Other): standard care
  Interventions: Other: Standard care
- 2 individualized PSP (Experimental): individualized patient support program
  Interventions: Other: individualized patient support program

INTERVENTIONS:
Other: individualized patient support program — individualized patient support with compliance supporting tools
  Arms: 2 individualized PSP
Other: Standard care
  Arms: 1 standard care

SUMMARY:
A 6 months prospective, randomized, multicenter, controlled, parallel-group, open-label study in RRMS patients to assess the impact of an individualized patient support program (PSP) on treatment satisfaction and to evaluate whether this individualized support improves satisfaction and with it adherence to medication compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this trial have to fulfill all of the following criteria:

1. Written informed consent from patients capable of giving or withholding full informed consent must be obtained before any assessment is performed.
2. Male or female subjects aged 18 - 65 years.
3. Subjects with relapsing remitting MS defined by 2010 revised McDonald criteria.
4. Patients with Expanded Disability Status Scale (EDSS) score of 0-6.5.
5. Patients under Fingolimod Therapy, according to German label, for at least 6 months at Study Visit 1 (Day 1).

Exclusion Criteria:

Patients fulfilling any of the following criteria are not eligible for inclusion in this study:

1. Patients, who are registered in any patient support program (e.g. Extracare)
2. Patients with any relevant medically unstable condition, as assessed by the primary treating physician at each site.
3. Any severe disability or clinical impairment that can prevent the patient to meet all study requirements at the investigator's discretion
4. History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin
5. Patients who have received an investigational drug (excluding Fingolimod) or therapy within 90 days or 5 half-lives prior to screening, whichever is longer.
6. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive pregnancy test (serum)
7. Women of childbearing potential unwilling to use contraceptive precautions throughout the study (see section 7.13.6 for details).
8. Simultaneous participation in another clinical trial.

Patients, who have already been randomized into this trial earlier must not be included a second time.

Study personnel or first degree relatives of investigator(s) must not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
change in treatment satisfaction (TSQM-9) from baseline to month 6 | 6 months
  To evaluate the effect of an individualized patient support program vs. a standard patient support program on treatment satisfaction, measured by a treatment satisfaction questionnaire (TSQM-9) in Fingolimod-treated patients with relapsing-remitting multiple sclerosis over 6 months.

SECONDARY OUTCOMES:
change in Modified Morisky Scale score from baseline to month 6 | 6 months
  To evaluate the effect of an individualized patient support program vs. standard care on therapy adherence, measured by an adherence questionnaire (Modified Morisky Scale) in Fingolimod-treated patients with relapsing-remitting multiple sclerosis over 6 months.
quantification of therapy adherence (pill-count) over 6 months | 6 months
  To evaluate the effect of an individualized patient support program vs. standard care on therapy adherence, measured by pill-count in Fingolimod-treated patients with relapsing-remitting multiple sclerosis over 6 months.
change in mFIS score from baseline to month 6 | 6 months
  To evaluate the effect of an individualized patient support program vs. standard care on fatigue, measured by mFIS in Fingolimod-treated patients with relapsing-remitting multiple sclerosis over 6 months.
change in BDI from baseline to month 6 | 6 months
  To evaluate the effect of an individualized patient support program vs. standard care on depression parameters, measured by the Beck depression inventory (BDI) in Fingolimod-treated patients with relapsing-remitting multiple sclerosis over 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals